CLINICAL TRIAL: NCT03035539
Title: Rehabilitation of Patients With Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Albert Marni Joensen, MD, PhD, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-20120002
Record Dates: First submitted 2012-07-13; First posted 2017-01-30 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Atrial Fibrillation
Keywords: Rehabilitation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Physiotherapists evaluating the physical capacity were masked.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard treatment (Active Comparator): Standard treatment after randomization
  Interventions: Other: Standard treatment
- Cardiac Rehabilitation (Experimental): The rehabilitation programme includes education, physical exercise, optimisation of the medical treatment, and discussion of implications for the daily life of each participant.
  Interventions: Other: Cardiac rehabilitation

INTERVENTIONS:
Other: Cardiac rehabilitation — AF specific cardiac rehabilitation Group education 1 hour each week for 3 months Physical training 1 hour each week for 3 months with physiotherapist
  Arms: Cardiac Rehabilitation
Other: Standard treatment — Standard treatment
  Arms: Standard treatment

SUMMARY:
The purpose of this study is to investigate whether a rehabilitation programme can improve the quality of life and reduce morbidity in patients with atrial fibrillation.

In addition, the study will map the economic costs and benefits of such a rehabilitation programme.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most frequent cardiac arrhythmia and is the cause of increased morbidity, mortality and socioeconomic costs.

Research conducted in recent years suggests that various pharmacological therapies and life style changes may affect the structural remodelling, thereby preventing the incidence of AF (primary prophylaxis) and a progression of the disease (secondary prophylaxis). These therapies, known as upstream therapy, include ace inhibitors/angiotensin II inhibitors, statins, the intake of n-3 polyunsaturated fatty acids and moderate physical exercise.

Furthermore, an important part of the treatment is to alleviate patients' symptoms, reduce the risk of thromboembolic complications and teach the patients to live with a chronic paroxysmal disease. Today, well-established pharmacological therapies are available, but there is only sparse knowledge of the effect of non-pharmacological therapies, how patients obtain information on the disease, how they learn how to cope with their symptoms, and how they relate to the uncertainty as to when they will experience the next symptom-producing attack of AF.

Cardiac rehabilitation is a collective term for the aftercare of patients with chronic heart failure. Cardiac rehabilitation is a cross-functional approach with participation of physicians, nurses, dieticians and smoking cessation instructors and is performed under the supervision of a cardiac specialist.

Cardiac rehabilitation includes: individually designed treatment plan, offer of patient information and education, support for smoking cessation, support for diet change, psychosocial support, optimisation of medical treatment and risk factor control, advice on physical exercise and maintenance of targets.

There is strong evidence that rehabilitation has a beneficial effect on the quality of life, but also on morbidity and mortality from other heart diseases than AF.

Currently, patients with the diagnosis of AF are not offered a rehabilitation programme, and there is sparse knowledge of the effect of rehabilitation on patients' quality of life and morbidity.

It is therefore of vital importance to develop and implement a rehabilitation programme aimed at improving the quality of life of patients with AF and, possibly, preventing admissions and the development of AF.

All participants are examined by exercise ECG to assess their maximum physical capacity (estimated oxygen uptake), Six-minute-walk test and Five-repetition-sit-to-stand test at inclusion and after 3 and 6 months.

At inclusion and at the end of the study each participant is to complete the QOL questionnaire, AF-QOL-18 and AFEQT, and questionnaire on lifestyle, heart symptoms, risk factors, medical treatment and sickness absence, if any, visits to own GP due to AFLI and hospital admissions.

The resource consumption for each individual participant is regularly recorded. Instructors and physiotherapists record their total time consumption (preparation and confrontation time) as well as patients' total time consumption (transportation and time for education/exercise. Furthermore, travel expenses in relation to rehabilitation are recorded. In addition the patients are to complete a questionnaire on lifestyle (Euroqol eq-5d) at inclusion and after 1, 3, 6 and twelve months, respectively, for use in the cost-benefit analysis. Data on visits to own GP are collected from the Danish Health Insurance Registry at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal or persistent atrial fibrillation
* Signed informed consent

Exclusion Criteria:

* Participating in other clinical trials
* Participating in other cardiac rehabilitation
* Atrial fibrillation secondary to electrolyte imbalance, thyroid disease, reversible or non-cardiac cause
* Other cardiac disease
* Unable to complete physical training

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-05; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in Quality of life measurement (AFEQT score) from baseline to 3, 6 and 12 months | Inclusion and at 3, 6 and 12 months
Change in Quality of life measurement (AF-QoL 18 score) from baseline to 3, 6 and 12 months | Inclusion and at 3, 6 and 12 months
Change in Quality of life measurement (GAD7 score) from baseline to 3, 6 and 12 months | Inclusion and at 3, 6 and 12 months
Change in Quality of life measurement (PHQ-9 score) from baseline to 3, 6 and 12 months | Inclusion and at 3, 6 and 12 months

SECONDARY OUTCOMES:
Morbidity | 12 months follow-up
Health Economics (Cost-effectiveness analysis) | 12 months follow-up
  Evaluated by
  - EQ-5
Change in maximum exercise capacity (calculated oxygen uptake) from baseline to 3 and 6 months | Inclusion and at 3 and 6 months follow up
Change in 6 minute walk test from baseline to 3 and 6 months | Inclusion and at 3 and 6 months follow up
Change in 5-repetition-sit-to-stand-test from baseline to 3 and 6 months | Inclusion and at 3 and 6 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Albert Marni Joensen, MD, PhD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] European Heart Rhythm Association; European Association for Cardio-Thoracic Surgery; Camm AJ, Kirchhof P, Lip GY, Schotten U, Savelieva I, Ernst S, Van Gelder IC, Al-Attar N, Hindricks G, Prendergast B, Heidbuchel H, Alfieri O, Angelini A, Atar D, Colonna P, De Caterina R, De Sutter J, Goette A, Gorenek B, Heldal M, Hohloser SH, Kolh P, Le Heuzey JY, Ponikowski P, Rutten FH. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). Eur Heart J. 2010 Oct;31(19):2369-429. doi: 10.1093/eurheartj/ehq278. Epub 2010 Aug 29. No abstract available. PMID 20802247
- [Background] Stewart S, Hart CL, Hole DJ, McMurray JJ. A population-based study of the long-term risks associated with atrial fibrillation: 20-year follow-up of the Renfrew/Paisley study. Am J Med. 2002 Oct 1;113(5):359-64. doi: 10.1016/s0002-9343(02)01236-6. PMID 12401529
- [Background] Hylek EM, Go AS, Chang Y, Jensvold NG, Henault LE, Selby JV, Singer DE. Effect of intensity of oral anticoagulation on stroke severity and mortality in atrial fibrillation. N Engl J Med. 2003 Sep 11;349(11):1019-26. doi: 10.1056/NEJMoa022913. PMID 12968085
- [Background] Savelieva I, Kourliouros A, Camm J. Primary and secondary prevention of atrial fibrillation with statins and polyunsaturated fatty acids: review of evidence and clinical relevance. Naunyn Schmiedebergs Arch Pharmacol. 2010 Mar;381(3):1-13. doi: 10.1007/s00210-009-0468-y. Epub 2009 Nov 25. PMID 19937318
- [Background] Anand K, Mooss AN, Hee TT, Mohiuddin SM. Meta-analysis: inhibition of renin-angiotensin system prevents new-onset atrial fibrillation. Am Heart J. 2006 Aug;152(2):217-22. doi: 10.1016/j.ahj.2006.01.007. PMID 16875900
- [Background] Aizer A, Gaziano JM, Cook NR, Manson JE, Buring JE, Albert CM. Relation of vigorous exercise to risk of atrial fibrillation. Am J Cardiol. 2009 Jun 1;103(11):1572-7. doi: 10.1016/j.amjcard.2009.01.374. Epub 2009 Apr 22. PMID 19463518
- [Background] Mozaffarian D, Furberg CD, Psaty BM, Siscovick D. Physical activity and incidence of atrial fibrillation in older adults: the cardiovascular health study. Circulation. 2008 Aug 19;118(8):800-7. doi: 10.1161/CIRCULATIONAHA.108.785626. Epub 2008 Aug 4. PMID 18678768
- [Background] Mont L, Sambola A, Brugada J, Vacca M, Marrugat J, Elosua R, Pare C, Azqueta M, Sanz G. Long-lasting sport practice and lone atrial fibrillation. Eur Heart J. 2002 Mar;23(6):477-82. doi: 10.1053/euhj.2001.2802. PMID 11863350
- [Background] Hegbom F, Sire S, Heldal M, Orning OM, Stavem K, Gjesdal K. Short-term exercise training in patients with chronic atrial fibrillation: effects on exercise capacity, AV conduction, and quality of life. J Cardiopulm Rehabil. 2006 Jan-Feb;26(1):24-9. doi: 10.1097/00008483-200601000-00005. PMID 16617223
- [Background] Osbak PS, Mourier M, Kjaer A, Henriksen JH, Kofoed KF, Jensen GB. A randomized study of the effects of exercise training on patients with atrial fibrillation. Am Heart J. 2011 Dec;162(6):1080-7. doi: 10.1016/j.ahj.2011.09.013. PMID 22137082
- [Background] European Association of Cardiovascular Prevention and Rehabilitation Committee for Science Guidelines; EACPR; Corra U, Piepoli MF, Carre F, Heuschmann P, Hoffmann U, Verschuren M, Halcox J; Document Reviewers; Giannuzzi P, Saner H, Wood D, Piepoli MF, Corra U, Benzer W, Bjarnason-Wehrens B, Dendale P, Gaita D, McGee H, Mendes M, Niebauer J, Zwisler AD, Schmid JP. Secondary prevention through cardiac rehabilitation: physical activity counselling and exercise training: key components of the position paper from the Cardiac Rehabilitation Section of the European Association of Cardiovascular Prevention and Rehabilitation. Eur Heart J. 2010 Aug;31(16):1967-74. doi: 10.1093/eurheartj/ehq236. Epub 2010 Jul 19. PMID 20643803
- [Background] Du H, Newton PJ, Salamonson Y, Carrieri-Kohlman VL, Davidson PM. A review of the six-minute walk test: its implication as a self-administered assessment tool. Eur J Cardiovasc Nurs. 2009 Mar;8(1):2-8. doi: 10.1016/j.ejcnurse.2008.07.001. Epub 2008 Aug 9. PMID 18694656
- [Background] Bohannon RW. Test-retest reliability of the five-repetition sit-to-stand test: a systematic review of the literature involving adults. J Strength Cond Res. 2011 Nov;25(11):3205-7. doi: 10.1519/JSC.0b013e318234e59f. PMID 21904240
- [Background] Arribas F, Ormaetxe JM, Peinado R, Perulero N, Ramirez P, Badia X. Validation of the AF-QoL, a disease-specific quality of life questionnaire for patients with atrial fibrillation. Europace. 2010 Mar;12(3):364-70. doi: 10.1093/europace/eup421. Epub 2010 Jan 6. PMID 20056594
- [Background] Spertus J, Dorian P, Bubien R, Lewis S, Godejohn D, Reynolds MR, Lakkireddy DR, Wimmer AP, Bhandari A, Burk C. Development and validation of the Atrial Fibrillation Effect on QualiTy-of-Life (AFEQT) Questionnaire in patients with atrial fibrillation. Circ Arrhythm Electrophysiol. 2011 Feb;4(1):15-25. doi: 10.1161/CIRCEP.110.958033. Epub 2010 Dec 15. PMID 21160035
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Goldsmith KA, Dyer MT, Buxton MJ, Sharples LD. Mapping of the EQ-5D index from clinical outcome measures and demographic variables in patients with coronary heart disease. Health Qual Life Outcomes. 2010 Jun 4;8:54. doi: 10.1186/1477-7525-8-54. PMID 20525323
- [Background] Dyer MT, Goldsmith KA, Sharples LS, Buxton MJ. A review of health utilities using the EQ-5D in studies of cardiovascular disease. Health Qual Life Outcomes. 2010 Jan 28;8:13. doi: 10.1186/1477-7525-8-13. PMID 20109189
- [Background] Brazier JE, Yang Y, Tsuchiya A, Rowen DL. A review of studies mapping (or cross walking) non-preference based measures of health to generic preference-based measures. Eur J Health Econ. 2010 Apr;11(2):215-25. doi: 10.1007/s10198-009-0168-z. Epub 2009 Jul 8. PMID 19585162
- [Background] Badia X, Arribas F, Ormaetxe JM, Peinado R, de Los Terreros MS. Development of a questionnaire to measure health-related quality of life (HRQoL) in patients with atrial fibrillation (AF-QoL). Health Qual Life Outcomes. 2007 Jul 4;5:37. doi: 10.1186/1477-7525-5-37. PMID 17610734
- [Background] Wittrup-Jensen KU, Lauridsen J, Gudex C, Pedersen KM. Generation of a Danish TTO value set for EQ-5D health states. Scand J Public Health. 2009 Jul;37(5):459-66. doi: 10.1177/1403494809105287. Epub 2009 May 1. PMID 19411320